CLINICAL TRIAL: NCT02559960
Title: Post-marketing Safety Surveillance of Breviscapine Powder-Injection : a Registry Study
Status: Suspended | Type: Observational
Sponsor: Zhong Wang (Other)
Responsible Party: Sponsor-Investigator, Zhong Wang, Dr, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: Dengzhan-V1.0
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Adverse Drug Event; Adverse Drug Reaction; Chinese Medicine; Anaphylactic Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breviscapine Powder-Injection: Breviscapine Powder-Injection will be given to the patients, and the investigators will record all the information including ADR, application of Breviscapine Powder-Injection and the combined medications, etc.
  Interventions: Drug: Breviscapine Powder-Injection

INTERVENTIONS:
Drug: Breviscapine Powder-Injection — Patients will be given Breviscapine Powder-Injection according to their disease condition in the real world. The investigator only can record the information on the usage of the drug and the relevant medications without any interventions.
  Other Names: Zhusheyong Deng-zhan-hua-su

SUMMARY:
This registry aims to monitor the safety of Breviscapine Powder-Injection and to identify the potential risk factors for the adverse drug reactions.

DETAILED DESCRIPTION:
Breviscapine Powder-Injection is a kind of natural compound injection with high purity of Scutellarin-Na (over 98%). It's a popular drug for ischemic diseases, as cerebral ischemic stroke, coronary heart disease or angor pectoris. However, more and more case reports about the adverse drug events of Chinese medicine injections extracted from Dengzhanhua (herba erigernotis) (Breviscapine is one of the most common compounds in it) have been reported in recent 10 years. Therefore, this registry of Breviscapine Powder-Injection aims to monitor the safety of Breviscapine Powder-Injection and to identify the potential risk factors for the adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use Breviscapine Powder-Injection in the monitoring departments of centain hospitals

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who use Breviscapine Powder-Injection in the monitoring departments of centain hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of anaphylactic reaction to Breviscapine Powder-Injection | 1 years

SECONDARY OUTCOMES:
The incidence of severe adverse events (SAEs) to Breviscapine Powder-Injection | 1 years
The incidence of new SAEs to Breviscapine Powder-Injection | 1 years
The incidence of adverse drug events (ADEs) to Breviscapine Powder-Injection | 1 years
The incidence of new ADEs to Breviscapine Powder-Injection | 1 years
The effective rate of Breviscapine Powder-Injection | 1 years
  The proportion of the patients whose drug effect is considered as "effective" by investigator.
The patient satisfaction rate for the therapy of Breviscapine Powder-Injection | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, M.D., Study Director — China Academy of Chinese Medical Sciences; Xin-zhi Wang, Principal Investigator — The First Hospital of Henan College of Traditional Chinese Medicine
Locations (15):
- China (15):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The People's Hospital of Zuanjiang District, Chongqing City, Chongqing, Chongqing Municipality
  - Mudanjiang City Second People's Hospital, Mudanjiang, Heilongjiang
  - People's Hospital of Jun County, Hebi, Henan
  - People's Hospital of Changge City, Xuchang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou Second Hospital, Zhengzhou, Henan
  - The First Hospital of Henan College of Traditional Chinese Medicine, Zhengzhou, Henan
  - Zaozhuang Hospital of T.C.M, Zaozhuang, Shandong
  - Shandong Energy Zaozhuang Mining Group Center Hospital, Zaozhuang, Shandong
  - Shanxi Provincial Hospital of Traditional Chinese Medicine, Taiyuan, Shanxi
  - Changzheng Hospital of Tianjin City, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Red Cross Hosptal of Yunnan, Kunming, Yunnan
  - First Affilicated Hospital of Kunming Medical University, Kunming, Yunnan